CLINICAL TRIAL: NCT05648006
Title: A Prospective, Multicenter, Open, Randomized Controlled Phase II Clinical Study Evaluating Recombinant Oncolytic HSV2（OH2）Therapeutic Injecta(Vero Cell) for Human Use(rHSV2hGM-CSF) in Combination With Capecitabine for First-line Maintenance Therapy in Advanced Colorectal Cancer
Brief Title: First-line Maintenance of OH2 Injection for Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategy adjustment
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-010
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Advanced Colorectal Carcinoma
Keywords: Oncolytic Virus
MeSH Terms: interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OH2+Capecitabine (Experimental): OH2: 10^7 CCID50/mL intratumoral injection, once every 2 weeks; Capecitabine: 1000 mg/m2, orally administered twice a day, D1 to D14, repeated every 3 weeks
  Interventions: Biological: OH2; Drug: Capecitabine
- Capecitabine/Capecitabine+Bevacizumab (Active Comparator): Capecitabine: 1000 mg/m2, orally administered twice a day, D1 to D14, repeated every 3 weeks Bevacizumab: 7.5 mg/kg, intravenously, once every 3 weeks.
  Interventions: Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Biological: OH2 — Oncolytic Type 2 Herpes Simplex Virus
  Arms: OH2+Capecitabine
Drug: Capecitabine — 1000 mg/m2, orally administered twice a day, D1 to D14, repeated every 3 weeks
Drug: Bevacizumab — Bevacizumab: 7.5 mg/kg, intravenously, once every 3 weeks.
  Arms: Capecitabine/Capecitabine+Bevacizumab

SUMMARY:
This is a prospective, multicenter, open, randomized controlled Phase II clinical study to evaluate the efficacy and safety of intratumoral injection of OH2 combined with capecitabine for first-line maintenance of advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (including boundary values), male or female;
2. Patients with advanced colorectal adenocarcinoma (Stage IV) with a definite histological or cytological diagnosis;
3. Partial response (PR) or stable disease (SD) was evaluated in advanced colorectal cancer patients after 16 to 24 weeks of first-line treatment with fluorouracil-based chemotherapy combined with or without targeted drugs, and before the last chemotherapy to trial drug administration;
4. The physical status score of the Eastern Oncology Consortium (ECOG) was 0~1;
5. Have at least one measurable or evaluable lesion according to RECIST 1.1;
6. There are lesions suitable for intratumoral injection;
7. At least 2 weeks and no more than 4 weeks after the end of the last first-line chemotherapy;
8. Expected survival ≥12 weeks;
9. Patients with asymptomatic BMS after treatment who are free of disease progression by computed tomography (CT) or magnetic resonance imaging (MRI), stable for at least 12 weeks and without steroid medication for at least 4 weeks;
10. Laboratory examination (no blood transfusion or use of blood products, no correction therapy with granulocyte colony stimulating factor or other hematopoietic stimulating factor within 14 days prior to the first dose) :

    1. WBC≥3.0×109/L, ANC≥1.5×109/L, PLT≥100×109/L, Hb≥90 g/L;
    2. Serum creatinine ≤1.5×ULN;
    3. TBIL≤1.5×ULN;
    4. ALT and AST≤2.5×ULN; Patients with liver metastasis ≤5×ULN;
    5. Normal coagulation: International normalized ratio INR≤1.5×ULN or prothrombin time (PT, APTT) ≤1.5×ULN;
11. For patients with herpes, it takes 3 months after the herpes subsides;
12. I have fully understood the research and voluntarily signed the informed consent, and I expect good compliance;
13. For women of childbearing age, the blood pregnancy test must be negative within 7 days before the first medication;
14. The use of at least one medically approved contraceptive method (e.g. surgical sterilization, oral contraceptives, intrauterine devices, controlled sexual desire or barrier contraception combined with spermicide) by fertile women and men with a partner of a woman of reproductive age for at least six months from the signing of the informed consent form until the last trial drug treatment.

Exclusion Criteria:

1. Patients who plan to undergo radical excision of metastatic lesions；
2. Unrelieved intestinal obstruction or malabsorption syndrome;
3. Adverse reactions caused by first-line chemotherapy drugs did not recover to ≤ grade 1 before randomization (except hair loss and peripheral neurotoxicity less than or equal to grade 2);
4. Cardiovascular disease meets one of the following criteria: Congestive heart failure with ≥NYHA Level III heart function; Severe arrhythmias requiring medical treatment; Acute myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass grafting, or stenting within 6 months prior to initial administration; Left ventricular ejection fraction (LVEF) <50%; Adjusted QTc interval (Fridericia formula correction) >450 ms for men and >470 ms for women, or risk factors for tip twisting ventricular tachycardia such as clinically significant hypokalemia as determined by the investigator, a family history of long QT syndrome, or a family history of arrhythmia (such as pre-excited syndrome); High blood pressure that is not effectively controlled;
5. Patients had active infection or unexplained fever >38.5℃ during screening or before initial administration;
6. Patients with congenital or acquired immune deficiency (such as HIV infection), syphilis antibody positive and syphilis rapid plasma reactin-positive, active hepatitis (hepatitis B: HBsAg positive and HBV DNA≥2000 IU/mL; Hepatitis C: HCV antibody positive and HCV virus copy number > upper limit of normal);
7. Had received or was receiving or still required to receive other experimental agents or antiviral therapy within 4 weeks before randomization (hepatitis B patients were treated with entecavir, tenofovir fumarate dipifurofurl, adefovir dipivoxil sustainably);
8. Participated in other clinical studies within 4 weeks prior to randomization;
9. Known to be allergic to the test drug or its active ingredients or excipients, or severely allergic;
10. A known history of psychotropic substance abuse, alcohol or drug abuse;
11. Patients who developed other malignant tumors within 5 years prior to inclusion, except for cervical carcinoma in situ, low-risk gastrointestinal stromal tumor, in situ or early stage breast cancer, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and papillary carcinoma of the thyroid, which were effectively resected and required no further antitumor therapy and had a recurrence survival rate of more than 70% in 5 years;
12. Patients with active autoimmune disease or a history of autoimmune disease that may recur, but patients with the following diseases are not excluded and can be further screened:

    1. Type 1 diabetes
    2. Hypothyroidism (if controlled with hormone replacement therapy alone)
    3. Controlled celiac disease
    4. Skin diseases that do not require systemic treatment (e.g. vitiligo, psoriasis, hair loss)
13. Patients for any condition requiring systemic therapy with glucocorticoids (prednisone >10 mg/ day or equivalent dose of the same drug) or other immunosuppressant within 14 days prior to the administration of the investigational drug, but who are currently or previously on any of the following steroid regimens may be enrolled:

    1. Epinephrine substitute steroid (prednisone ≤10 mg/ day or equivalent dose of similar drugs)
    2. Systemic absorption of minimal amounts of local, ocular, intra-articular, intranasal or inhaled corticosteroids
    3. Prophylactic short-term (≤7 days) use of corticosteroids (e.g., allergy to contrast media) or to treat non-autoimmune conditions (e.g., delayed hypersensitivity caused by contact allergens)
14. Patients with grade 2 or above radiation pneumonia during previous antitumor therapy, or pulmonary diseases such as pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severe impairment of lung function;
15. Pleural effusion or ascites with clinical symptoms requiring repeated drainage (≥1 time/month);
16. Other researchers did not consider it appropriate to participate in this study.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Time after treatment to clinical and radiographic disease progression will be evaluated.

SECONDARY OUTCOMES:
Durable response rate (DRR) | 2 years
  objective response lasting continuously 6 months
Overall survival (OS) | 2 years
  The overall survival for each patient receiving treatment will be calculated.
Objective response rate (ORR) | 2 years
  Determination of the ORR will be calculated based on the proportion of patients achieving CR or PR using the RECIST v1.1 and iRECIST as assessed by investigators.
Disease control rate (DCR) | 2 years
  DCR will be calculated based on the proportion of patients achieving CR, PR, or who have SD at least 6 weeks after receiving first dose of study treatment.
Duration of response (DoR) | 2 years
  DOR will be calculated from the time of initial response (CR or PR) documentation to the time of progressive disease (PD). If a subject who had CR or PR dies without the evidence of disease progression, the case will be censored at the time point of death when analyzing DOR
Immune-progression-free survival (iPFS) | 2 years
  Time after treatment to disease progression using the iRECIST will be evaluated.
Toxicity by CTCAE v5.0 | 2 years
  Safety assessments should be conducted for all subjects who received treatment at least once. Adverse events will be graded according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China